CLINICAL TRIAL: NCT00061750
Title: A Randomized, Comparative, Open Label Phase III Trial on Efficacy & Safety of Long-term Treatment With ICL670 Compared to Deferoxamine in Beta-thalassemia Patients With Transfusional Hemosiderosis
Brief Title: Safety & Efficacy of ICL670 vs. Deferoxamine in Beta-thalassemia Patients With Iron Overload Due to Blood Transfusions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CICL670A0107
Record Dates: First submitted 2003-06-03; First posted 2003-06-04 (Estimated); Last update posted 2012-04-19 (Estimated); Status verified 2012-04

CONDITIONS: Beta-Thalassemia
Keywords: Thalassemia, iron overload, deferoxamine, hemosiderosis
MeSH Terms: conditions — beta-Thalassemia; Thalassemia; Iron Overload; Hemosiderosis | interventions — Deferasirox; Deferoxamine

ARMS (2):
- ICL670 (Experimental)
  Interventions: Drug: ICL670
- Deferoxamine (Active Comparator)
  Interventions: Drug: deferoxamine

INTERVENTIONS:
Drug: ICL670
  Other Names: Deferasirox
  Arms: ICL670
Drug: deferoxamine
  Arms: Deferoxamine

SUMMARY:
The purpose of this study is to deterimine if the new orally active iron chelator, ICL670, is as effective and as safe as deferoxamine in preventing accumulation of iron in the body while a patient is undergoing repeated blood transfusions.

DETAILED DESCRIPTION:
Patients who require repeated blood transfusions to live accumulate iron in the body as blood cells contain iron and there is no natural body mechanism to eliminate it. After a while the iron levels get high enough to be toxic to the body. The current therapy of choice is deferoxamine, which does a good job of removing excess iron, but is difficult to administer. Deferoxamine requires subcutaneous (under the skin) infusions over 4 to 8 hours nightly 3 to 7 nights per week. In addition to the need to wear an infusion pump nightly, adverse reactions around the site of the injection are frequent.

ELIGIBILITY:
Inclusion Criteria:

* Beta-thalassemia patients already treated with or suitable for treatment with deferoxamine 20 to 40 mg/kg/day
* Liver iron content greater than 2 mg iron/g dw as measured by liver biopsy
* Need for regular transfusions 8 or more times per year

Exclusion Criteria:

* Non-transfusional iron overload or transfusion-dependent anemias other than beta-thalassemia.
* Documented toxicity to deferoxamine
* Elevated liver enzymes in the year preceeding enrollment
* Active hepatitis B or hepatitis C
* HIV seropositivity
* Elevated serum creatinine or significant proteinuria
* History of nephrotic syndrome
* Uncontrolled systemic hypertension
* Fever and other signs/symptoms of infection within 10 days prior to start of the study
* Presence of clinically relevant cataract or previous history of clinically relevant ocular toxicity related to iron chelation
* Second or third degree AV block, clinically relevant Q-T interval prolongation, or patients requiring digoxin or other drugs that prolong the Q-T interval
* Diseases (cardiovascular, renal, hepatic, etc.)that would prevent the patient from undergoing any of the treatment options
* Psychiatric or additive disorders that would prevent the patient from giving informed consent
* History of drug or alcohol abuse within the 12 months prior to the study
* Pregnant or breast feeding patients
* Patients treated with systemic investigational drugs within 4 weeks or topical investigational drugs within 7 days before the start of the study
* Any surgical or medical condition that might significantly alter the absorption, distribution, metabolism or excretion of any drug, such as gastrointestinal disease or major surgery, renal disease, difficulty voiding or urinary obstruction, or impaired pancreatic function.
* Non-compliant or unreliable patients.
* Patients unable to undergo any study procedures such as the hearing or eye tests, or the liver echocardiography.
* Inability to undergo a liver biopsy.
* Patients that would need a dose of ICL670 less than 125 mg per day.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 595 (Actual)
Dates: Start 2003-05; Primary Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
Demonstrate non-inferiority to deferoxamine in its effects on liver iron content (LIC)

SECONDARY OUTCOMES:
Evaluate tolerability profile
Estimate absolute and relative change of LIC and Total body iron excretion
Evaluation relationship between LIC and potential surrogate markers
Evaluate the relationship between pharmacokinetics, pharmacodynamics and safety variable

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- United States (7):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Children's Hospital Oakland, Oakland, California
  - Stanford Hospital, Stanford, California
  - Children's Memorial Hospital, Chicago, Illinois
  - Children's Hospital Boston, Boston, Massachusetts
  - Weill Medical College of Cornell University, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Padhani ZA, Gangwani MK, Sadaf A, Hasan B, Colan S, Alvi N, Das JK. Calcium channel blockers for preventing cardiomyopathy due to iron overload in people with transfusion-dependent beta thalassaemia. Cochrane Database Syst Rev. 2023 Nov 17;11(11):CD011626. doi: 10.1002/14651858.CD011626.pub3. PMID 37975597
- [Derived] Cohen AR, Glimm E, Porter JB. Effect of transfusional iron intake on response to chelation therapy in beta-thalassemia major. Blood. 2008 Jan 15;111(2):583-7. doi: 10.1182/blood-2007-08-109306. Epub 2007 Oct 19. PMID 17951527